CLINICAL TRIAL: NCT01182727
Title: Salsalate for the Treatment of Insulin Resistance in People With Schizophrenia
Brief Title: Salsalate for Insulin Resistance in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00046612
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia; Insulin Resistance
Keywords: schizophrenia; salsalate; obesity
MeSH Terms: conditions — Schizophrenia; Insulin Resistance; Obesity | interventions — salicylsalicylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- salsalate (Experimental): Salsalate will be administered in two divided doses of 2grams in the morning and 2 grams in the evening. Salsalate will be administered for 6 weeks. If a participant is not able to tolerate the target dose of 4 grams per day then 500 mg reductions will be made in a stepwise fashion until a tolerated dose or a minimum dose of 2 grams per day is reached.
  Interventions: Drug: salsalate

INTERVENTIONS:
Drug: salsalate — Salsalate will be administered in 500 mg tablets. Salsalate will be administered in two divided doses of 2 grams in the morning and 2 grams in the evening. Salsalate will be administered for a total of 6 weeks. If a participant is not able to tolerate the target dose of 4 grams per day then 500 mg reductions will be made in a stepwise fashion until tolerated or a minimum dose of 2 grams per day is achieved.

SUMMARY:
Being obese is a common problem for people with schizophrenia. People with schizophrenia are more likely to be overweight compared to the general population. Being overweight is a major risk factor for developing type II diabetes. Approximately 15% of people with schizophrenia have type II diabetes. People with type II diabetes have problems with their body's insulin. Insulin is a hormone produced by the body to control blood sugar level. Obesity and type II diabetes are strong risk factors for heart disease. In type II diabetes the body does not respond to insulin correctly. Obesity, type II diabetes, and insulin resistance are all common states of inflammation. Inflammation is a reaction by the body to irritation, injury, or infection.

Salicylates are non-steroidal anti-inflammatory drugs. Aspirin is an example of a salicylate. These drugs work by decreasing the level of inflammation in the body. Salicylates have been shown to decrease inflammation and improve the body's response to insulin. Improving the body's response to insulin and decreasing inflammation could possibly reduce the risk of developing type II diabetes. Salicylates have been known for years to be effective for the treatment of diabetes. Salicylates increase the body's response to insulin causing blood sugar levels to decrease. Many salicylate drugs have side effects including stomach irritation and increased risk of bleeding. The drug for this study is called salsalate and is different from other salicylates. Salsalate has a lower bleeding risk than aspirin. Salsalate has been used to treat arthritis and has been shown to be safe.

There have been no studies using salsalate in people with schizophrenia. The purpose of this study is to gain experience in the use of salsalate in people with schizophrenia. The study would be a pilot study to obtain preliminary data. The study would be a 6-week study where everyone in the study would receive the drug salsalate. The participants in the study will have tests of baseline symptoms of schizophrenia, a physical exam, EKG (to check heart function), and a side effect checklist for possible side effects from salsalate. The study will also have some blood drawn to measure blood sugar levels, insulin levels, and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV TR diagnosis of schizophrenia or schizoaffective disorder
* Body Mass Index (BMI) greater than or equal to 27 kg/m2
* Participant will be judged to be clinically stable
* Participants will be treated with the same antipsychotic for at least 90 days and will have received a constant therapeutic dose for at least 20 days prior to study entry. There will not be any restriction on the type of antipsychotic with which the participant is treated.
* Participants must be judged competent to participate in the informed consent process and provide voluntary informed consent.

Exclusion Criteria:

* Individuals with aspirin allergy.
* Individuals with pre-existing tinnitus.
* Individual with anemia or thrombocytopenia.
* Individuals with ongoing infections.
* Individuals with history of autoimmune disease.
* Individuals with peptic ulcer disease or gastritis.
* Individuals with weight loss greater than 5% over the past 6 months.
* Individuals currently taking immunosuppressive drugs including corticosteroids.
* Individuals taking anti-diabetic agents.
* Individuals taking non-steroidal anti-inflammatory agents (other than low dose aspirin).
* Individuals with organic brain disorder; mental retardation; or medical conditions whose pathology or treatment would alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol.
* Pregnant females.
* Individuals who meet DSM-IV TR criteria for alcohol or substance dependence (except nicotine) within the last 6 months.
* Individuals who meet DSM-IV TR criteria for alcohol or substance abuse (except nicotine) within the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, MD, Principal Investigator — University of Maryland School of Medicine Maryland Psychiatric Research Center
Locations (2):
- United States (2):
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Maryland Psychiatric Research Center, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from August 2010 to August 2011 from multiple community mental health clinics.
Pre-assignment Details: Participants were withdrawn from the trial if they had abnormal lab values or were found to have a diagnosis of diabetes.
Period: Overall Study
Arm/Group | Salsalate
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Salsalate
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Side Effects of Salsalate
Description: This Measure is reporting the number of participants with side effects as reported on the Side Effect Checklist used to monitor common medication side effects.
Time Frame: 6 weeks
Population: All subjects who completed the study were analyzed.
Measure: Number; unit: participants
Arm/Group | Salsalate
Number analyzed (Participants) | 10
participants | 3

ADVERSE EVENTS:
Arm/Group | Salsalate
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No